CLINICAL TRIAL: NCT07053800
Title: A Single-Arm, Open-Label, Phase II Study to Determine the Safety and Efficacy of Obecabtagene Autoleucel (Obe-cel) in Participants With Severe, Refractory Systemic Lupus Erythematosus With Active Lupus Nephritis
Brief Title: Obe-cel in Severe, Refractory Systemic Lupus Erythematosus With Active Lupus Nephritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO1-SL2; 2024-519941-32 (EudraCT Number); 1011415 (Other: UK IRAS ID)
Record Dates: First submitted 2025-05-13; First posted 2025-07-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lupus Nephritis
Keywords: Systemic lupus erythematosus; Refractory systemic lupus erythematosus; Lupus nephritis; Obecabtagene autoleucel; Obe-cel
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Single-arm, single group assignment, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obe-cel (Experimental)
  Interventions: Biological: Obecabtagene autoleucel

INTERVENTIONS:
Biological: Obecabtagene autoleucel — Obecabtagene autoleucel (obe-cel) given as a single infusion
  Other Names: Obe-cel

SUMMARY:
This trial aims to find out if obe-cel gets rid of harmful B cells that contribute to systemic lupus erythematosus (SLE)/lupus nephritis (LN) when available treatments have not worked (refractory). The trial includes only 1 group of patients (single arm), including teenage and adult patients aged 12 to 65 years. The objective is to look for benefits of obe-cel in making signs of LN completely disappear (remission) at 6 months after treatment in patients with severe, active LN. The trial will also look for other benefits of obe-cel for up to 24 months after treatment, including the percentage of patients who respond to obe-cel treatment, SLE/LN activity, time to and length of remission, and quality of life. The trial will also assess how long obe-cel stays in the body and the safety of obe-cel.

DETAILED DESCRIPTION:
This is a Phase II study to determine the efficacy and safety of obe-cel in participants with severe, refractory SLE with active LN.

The study comprises 3 periods:

1. Screening Period: From Day -30 to Day of Enrolment
2. Treatment Period: From Day -8 to Day 1 - Patients will be evaluated to confirm eligibility for lymphodepletion, and thereafter receive lymphodepletion to enhance treatment efficacy and cluster of differentiation (CD)19 chimeric antigen receptor (CAR) T cell survival
3. Obe-cel Administration: If the participant's eligibility for receiving obe-cel infusion is confirmed, the participant is to receive a single obe-cel infusion on Day 1. From Day 1 to End of Study all participants will be followed up for efficacy and safety evaluation.

The objective is to look for benefits of obe cel in making signs of LN completely disappear (remission) at 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study or written informed consent signed by a legal guardian or representative
* Ability and willingness to adhere to protocol's Schedule of Activities and other requirements
* Participants must be 12 to 65 years of age inclusive at the time of signing the informed consent.
* Female Participants: - a female participant is eligible to participate if she is not pregnant or breastfeeding
* Diagnosis of SLE fulfilling the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) Classification Criteria for Systemic Lupus Erythematosus.
* Positive for at least 1 of the following autoantibodies: antinuclear antibodies (ANA), or anti-dsDNA or anti-Smith.
* Severe, Active SLE defined as:

  * Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score of ≥ 8 points AND
  * Severe active LN based on a renal biopsy obtained within 6 months prior to signing the informed consent form or during the screening period Class III, IV or V (V only in combination with class III or IV)
* Refractory SLE defined as failure to early lines of therapy and to Calcineurin inhibitors AND B cell-targeting agents

Exclusion Criteria:

* Any medications prohibited by the protocol.
* Prior treatment at any time with anti-CD19 therapy.
* More than 1 acute, severe lupus-related flare during screening that needs immediate treatment and/or makes the immunosuppressive washout impossible.
* Significant, likely irreversible organ damage related to SLE (e.g., end-stage renal disease) that in the opinion of the Investigator renders CD19 CAR T cell therapy unlikely to benefit the participant.
* History of primary antiphospholipid antibody syndrome.
* Active or uncontrolled fungal, bacterial, or viral infection
* History of malignant neoplasms unless disease free for at least 24 months.
* History of heart, lung, renal, liver transplant or hematopoietic stem cell transplant.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve complete renal response (CRR) at 6 months post-obe-cel infusion without rescue medications, among all participants who received obe-cel infusion | Month 6
  CRR is defined as change in
  * urine protein creatinine ratio (UPCR) and
  * estimated glomerular filtration rate (eGFR) without use of rescue medication

SECONDARY OUTCOMES:
Proportion of participants who achieve response according to Definition of Remission in SLE (DORIS) at 6 months post-obe-cel infusion, among all patients who received obe-cel infusion | Month 6
Proportion of participants with CRR. | Up to Month 24
  CRR is defined as change in UPCR and eGFR without use of rescue medication.
Time to CRR | Up to Month 24
  CRR is defined as change in UPCR and eGFR without use of rescue medication.
Duration of CRR. | Up to Month 24
  CRR is defined as change in UPCR and eGFR without use of rescue medication.
Proportion of participants with Partial Renal Response (PRR) | Up to Month 24
  PRR is defined as reduction in UPCR from baseline.
Remission over time as specified by DORIS. | Up to Month 24
Time to response, as specified by DORIS. | Up to Month 24
Remission over time, as specified by the definition of remission in Lupus Low Disease Activity State (LLDAS). | Up to Month 24
  Definition as specified by LLDAS
Time to remission and duration of remission, as specified by the definition of remission in LLDAS. | Up to Month 24
  Definition as specified by LLDAS
Time from obe-cel infusion to first disease flare according to definition of flare in Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI-2K Flare Index (SFI) | Up to Month 24
Changes from baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue | Up to Month 24
  Score range 0-52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life.
Changes from baseline in Disability Health Assessment Questionnaire - Disability Index (HAQ-DI). | Up to Month 24
  HAQ-DI instrument consists of 2 visual analog scales 1) the PtGA and 2) Pain scale. Both are scored from 0-100 with higher numbers representing worse perceived disease activity or overall health.
Changes from baseline in Short Form Health Survey (SF-36). | Up to Month 24
  The SF-36 score range is from 0 to 100. Higher scores indicate better perceived health, while lower scores indicate greater disability or poorer health. The SF-36 assesses eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health.
Changes from baseline in EuroQoL (EQ)-5 Dimension (D). | Up to Month 24
  EQ-5D index scores range from -0.59 to 1, where 1 is the best possible health state; EQ visual analog scale scores range from 0 to 100, where 100 is the best possible health state.
To evaluate safety of obe-cel | Up to Month 24
  Number of participants with Adverse events (AE).
Pharmacokinetics (PK) of CAR-T cells post obe-cel infusion - Maximum concentration (Cmax) | Up to Month 24
  Analysis of cells in peripheral blood at a range of time points.
Pharmacokinetics (PK) of CAR-T cells post obe-cel infusion - time to maximum concentration (Tmax) | Up to Month 24
  Analysis of cells in peripheral blood at a range of time points.
Pharmacokinetics (PK) of CAR-T cells post obe-cel infusion - last observed quantifiable concentration (Clast) | Up to Month 24
  Analysis of cells in peripheral blood at a range of time points.
Pharmacokinetics (PK) of CAR-T cells post obe-cel infusion - time to last observed quantifiable concentration (Tlast) | Up to Month 24
  Analysis of cells in peripheral blood at a range of time points.
Pharmacokinetics (PK) of CAR-T cells post obe-cel infusion - area under the curve (AUC) | Up to Month 24
  Analysis of cells in peripheral blood at a range of time points.
To evaluate pharmacodynamics (PD) of obe-cel | Up to Month 24
  Detection of B cells in the peripheral blood over time

IPD SHARING:
Plan to Share IPD: No